CLINICAL TRIAL: NCT02994628
Title: Influence of Bananas Varying in Carbohydrate and Phenolic Content on Exercise Performance and Recovery
Brief Title: Banana Cultivars and Exercise Performance and Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Appalachian State University (Other)
Collaborators: Dole Food Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 16-0071
Record Dates: First submitted 2015-11-24; First posted 2016-12-16 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2016-01

CONDITIONS: Inflammation
Keywords: oxidative stress; immune function; muscle damage; carbohydrate; polyphenols; cycling
MeSH Terms: conditions — Inflammation | interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Water (Active Comparator): Intervention, water and no banana carbohydrate: consume 3 ml/kg water every 15 min during 75 km cycling
  Interventions: Other: Water
- Mini banana (Experimental): Intervention, banana carbohydrate: ingest 0.2 g carbohydrate/kg body weight from Mini banana with 3 ml/kg water every 15 minutes during 75 km cycling
  Interventions: Other: Mini banana
- Cavendish banana (Experimental): Intervention, banana carbohydrate: ingest 0.2 g carbohydrate/kg body weight from Cavendish banana with 3 ml/kg water every 15 minutes during 75 km cycling
  Interventions: Other: Cavendish banana
- 6% sugar beverage (Experimental): Intervention: pure banana carbohydrate in sugar beverage; ingest 0.2 g carbohydrate/kg body weight from a 6% sugar beverage every 15 minutes during 75 km cycling (contains 60 grams sugar per liter using the same sugar profile found in Cavendish bananas)
  Interventions: Other: 6% sugar beverage

INTERVENTIONS:
Other: Water — Water only without carbohydrate
  Arms: Water
Other: Mini banana — Ingest mini banana containing higher phenolics and carbohydrate concentration
  Arms: Mini banana
Other: Cavendish banana — Ingest Cavendish banana (common banana)
  Arms: Cavendish banana
Other: 6% sugar beverage — Ingest 6% sugar beverage containing same glucose and fructose profile as banana
  Arms: 6% sugar beverage

SUMMARY:
In a previous study at the Appalachian State University (ASU) Human Performance Laboratory at the North Carolina Research Campus (NCRC), investigators showed that cyclists ingesting about one-half of a banana with water every 15 minutes cycled 75-km faster (5%) than with water alone. The polyphenols (i.e., chemicals in plants with health benefits) in the banana improved the capacity to counter oxidative stress, and the sugars lowered post-exercise inflammation. The cyclists reported some gastrointestinal discomfort, however, from the high volume of bananas consumed. Dole Foods, the sponsor of this study, has a banana collection that includes many different varieties, including the Mini banana that has a higher sugar (50%) and phenolic (63%) content than the typical banana (Cavendish) available in stores. Thus athletes should experience similar performance benefits from a smaller volume of Mini compared to Cavendish bananas, and reduced gastrointestinal symptoms. If study results are favorable, Dole Foods may market the Mini banana as the "sport" banana.

The purpose of this study is to compare ingestion of Mini and Cavendish bananas with an equicaloric, sugar-only beverage or water on 75-km cycling performance and post-exercise oxidative capacity and stress, inflammation, immune function, muscle damage and soreness, and gastrointestinal symptoms.

DETAILED DESCRIPTION:
The research procedures will be conducted at the Human Performance Laboratory (Room 1201, Plants for Human Health Institute Building, 600 Laureate Way), operated by Appalachian State University at the North Carolina Research Campus (NCRC) in Kannapolis, NC. Participants will come here for orientation/baseline testing and then 4 exercise test sessions (with each including two additional lab visits to provide 1- and 2-day 7:00 am recovery blood samples) (thus 13 total lab visits). The total amount of time participants will be asked to volunteer for this study is about 35 hours at the Human Performance Laboratory (over a 7 to 8-week period).

ORIENTATION AND BASELINE TESTING:

One to two weeks prior to the first 75-km cycling time trial, participants will report to the NCRC Human Performance Lab for orientation/baseline testing. Participants will be screened to verify "low risk" status for cardiovascular disease, and provide voluntary consent. Demographic and training histories will be acquired with questionnaires.

Participants will be tested for VO2max (i.e., maximal oxygen consumption) using the Lodi cycle ergometer. The purpose of the VO2max test is to determine maximum exercise capacity. The time commitment is about 30 to 60 minutes, and participants will wear exercise clothes and shoes that allow for free movement during vigorous exercise. Participants will be rested, well nourished, and hydrated for the test and avoid alcohol, caffeine, and tobacco 3 hours before the test. Participants will avoid significant exertion or exercise the day of testing and report any medication that are being used to the testing staff before the test. The test will begin with an exercise warm-up period of a few minutes, and then participants will pedal at progressively harder workloads. The test will continue until participants become fatigued and decide to stop, or other symptoms prohibit further exercise. Both leg tiredness and breathlessness are common sensations of the fatigue that participants may experience. During the test, participants will wear a facemask that allows exhaled air to be analyzed, and a chest strap for heart rate monitoring. Participants will communicate with the lab personnel during the test by the use of a perceived exertion chart to indicate how the exercise feels.

Percent body fat will be measured using the BodPod. Participants will sit inside the BodPod with a tight-fitting swim suit for about 10 minutes while body fat is calculated.

75-km CYCLING TIME TRIALS:

A. 3-day pre-75 km cycling preparation: During the 3-day period prior to each 75-km cycling trial, participants will taper exercise training (as if preparing for a race) and ingest a moderate-carbohydrate diet using a food list restricting high fat foods and visible fats. Participants will record all food and beverage intake during the 3-day period, with nutrient intake assessed using a computerized dietary analysis software system. Participants will bring the food log to each exercise lab session.

B. Testing procedures: Participants will come to the lab four times at 7:00 am in an overnight fasted state (at least 9 h with no food or beverage other than water) and complete 75-cycling time trials (at least two weeks apart) under four separate conditions (random order, crossover): Water only (WAT); Cavendish bananas and water (BAN); Mini bananas and water (SPORT-BAN); 6% carbohydrate beverage (SUGAR).

1. 7:00 am: A blood sample will be collected through a needle inserted into an arm vein (about 35 ml or 2.5 tablespoons). An ultrasound scan of the thigh muscle will be conducted to measure pre-exercise muscle glycogen levels. The side of the thigh will be scanned through a smooth probe attached to the General Electric LOGIQ-e ultrasound machine (GE Healthcare, Milwaukee, WI). Participants will lie on their backs with the skin over the thigh exposed. Three baseline scans will be obtained (each taking 10 seconds), just prior to the exercise test, and then this muscle will be scanned three times again following the exercise bout. A simple questionnaire will be used for to indicate muscle soreness (DOMS). Participants will complete a symptom log, which will include questions on digestive and mental health (heartburn, bloating, diarrhea, nausea, energy levels, ability to focus, etc.). Participants will indicate responses using a 12-point Likert scale, with 1 relating to "none at all", 6 "moderate", and 12 "very high".
2. 7:10 am: Ingest 5 ml/kg water alone (about 1.5 cups), or SUGAR beverage, or water (5 ml/kg) and BAN or SPORT-BAN (volume adjusted to provide 0.4 g carbohydrate per kilogram of body weight) (about two cups SUGAR beverage, one Cavendish banana, or 1.5 Mini bananas).
3. 7:30 am: Start 75-km cycling time trial. Participants are to complete the 75-km course as fast as possible.

   * Participants will use their own bicycles on CompuTrainer Pro Model 8001 trainers (RacerMate, Seattle, WA).
   * A mountainous 75-km course with moderate difficulty will be utilized using the CompuTrainer software system.
   * Heart rate and rating of perceived exertion (RPE) will be recorded every 30 minutes, and workload (watts) continuously monitored using the CompuTrainer MultiRider software system (version 3.0, RacerMate, Seattle, WA).
   * Oxygen consumption, carbon dioxide production, and ventilation will be measured using the Cosmed metabolic cart after 16 km and 55 km cycling (through a facemask similar to what occurred during baseline testing). Performance will be monitored throughout the 75-km cycling time trial using percentage of maximal watts to ensure that a full effort is being given.
   * Participants will consume 3 ml/kg water every 15 min (e.g., about one cup for a 75 kg cyclist).
   * Participants will ingest 0.2 g carbohydrate/kg body weight every 15 minutes of BAN, SPORT-BAN, or SUGAR beverage during the 75-km time trials. For a 75-kg cyclist, intake will be approximately 0.5 Cavendish banana, just under one Mini Banana, or one cup SUGAR beverage every 15 minutes. Bananas will be provided by Dole Foods at the appropriate ripening stage (equal to stage six). The SUGAR beverage will be prepared by Dole Foods, and will contain 60 grams sugar per liter using the same sugar profile found in Cavendish bananas.
   * No other beverage or food containing energy or nutrients will be allowed during the cycling time trials.
4. ~10:00-11:30 am: Immediate-post-exercise, 0.75-h, 1.5-h recovery blood samples; lunch

   * Blood samples will be taken from an arm vein immediately after completing the 75-km time trial, and then 0.75-h and 1.5-h post-exercise. Participants will be allowed to shower and change clothes in the facility.
   * An ultrasound scan for muscle glycogen levels will be conducted immediately post-exercise.
   * Immediately post-exercise, participants will complete the symptom log.
   * Participants will indicate muscle soreness using the DOMS questionnaire immediately post-exercise and 1.5-h post-exercise.
   * Participants will ingest no food or beverage other than water (7 ml/kg or about two cups during the 1.5 h post-exercise period).
   * Right after the 1.5-h recovery blood sample has been collected, participants will ingest a meal adjusted to 12 kcal/kg body weight. The meal will be prepared by Dole Foods and include grilled chicken, rice, corn, green beans, salt, and water.
5. ~11:30 am to 2:30 pm: 3-h and 4.5-h recovery

   * Additional blood samples will collected 3-h and 4.5-h post-exercise. During this time, participants will rest quietly in the lab.
   * The DOMS questionnaire will be administered 4.5-h post-exercise.
   * Participants will ingest no food or beverage other than water (7 ml/kg per hour).
   * At ~2:30 pm, participants will be allowed to leave the lab, and will be instructed to adhere to the food list requirements, and to keep exercise training intensity moderate with duration under 1.5 h per day.
6. 7:00 am: 21-h and 45-h Recovery samples (following two mornings) • Participants will return to the lab the following two mornings in an overnight fasted state at about 7:00 am (~21-h and 45-h after completing the 75-km time trial). Blood samples and responses to the DOMS questionnaire will be collected at both lab visits.

Blood samples will be analyzed for markers of muscle damage, inflammation and oxidative stress indicators (using blood levels and gene expression), and immune function. Stored samples will be measured for post-exercise shifts in hundreds of biochemicals using a special method called metabolomics, pending additional sponsor funding.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, with no known cardiovascular disease, diabetes, or cancer.
* Non-smoker.
* Regularly compete in road races (category 1 to 5) and/or capable of cycling 75 km in a laboratory setting (using own bicycles on CompuTrainer training systems).
* Agree to train normally, maintain weight, and avoid the regular use of large-dose vitamin and mineral supplements, herbs, and medications that influence inflammation and immune function (in particular, Advil, Motrin, aspirin and similar anti-inflammatory drugs) for the duration of the 7 to 8-week study. If in doubt, discuss supplement/medication use with the Research Manager.
* Categorized as "low risk" using the American College of Sports Medicine screening questionnaire.

Exclusion Criteria:

* Inability to comply with study requirements.
* Any other concurrent condition which, in the opinion of the primary investigator (PI), would preclude participation in this study or interfere with compliance.
* Current diagnosis of cardiovascular disease, diabetes, or cancer (except for non-melanoma skin cancer).

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-01-25 (Actual)

PRIMARY OUTCOMES:
Change in total plasma concentrations of inflammatory cytokines | Pre-exercise, and post-exercise (0, 0.75, 1.5, 3.0, 4.5, 21, 45 hours)
  Total plasma concentrations of five inflammatory cytokines [monocyte chemoattractant protein-1 (MCP-1), tumor necrosis factor alpha (TNFα), IL-6, IL-8, and IL-10] will be determined using an electrochemiluminescence based solid-phase sandwich immunoassay (Meso Scale Discovery, Gaithersburg,MD, USA).

SECONDARY OUTCOMES:
Change in concentration of serum myoglobin | Pre-exercise, and post-exercise (0, 0.75, 1.5, 3.0, 4.5, 21, 45 hours)
  muscle damage marker
Change in muscle concentration of glycogen | Pre-exercise, and post-exercise (0 hours)
  change in muscle glycogen using ultrasound
Change in self-reported gastrointestinal and mental symptoms from a short questionnaire | Pre-exercise, and post-exercise (0 hours)
  Gastrointestinal and mental symptoms, 1-12 Likert scale
Change in concentration of ferric reducing ability of plasma (FRAP) | Pre-exercise, and post-exercise (0, 0.75, 1.5, 3.0, 4.5, 21, 45 hours)
  total plasma antioxidant power
Change in plasma concentration of oxidized low density lipoprotein | Pre-exercise, and post-exercise (0, 0.75, 1.5, 3.0, 4.5, 21, 45 hours)
  oxidative stress
Change in blood natural killer cell activity | Pre-exercise, and post-exercise (0, 0.75, 1.5, 3.0, 4.5, 21, 45 hours)
  innate immune measure

CONTACTS AND LOCATIONS:
Overall Officials: David C. Nieman, DrPH, Principal Investigator — Appalachian State University, North Carolina Research Campus
Locations (1):
- Human Performance Lab, North Carolina Research Campus, Kannapolis, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared through the Human Metabolome Database (HMDB) or the Scripps Metabolite and Tandem MS Database (METLIN)], other public web sites, and publication in the scientific literature. We will cooperate in making available cloud-based access to the data and associated informatics components within the general scientific community.

REFERENCES:
- [Background] Nieman DC, Gillitt ND, Sha W, Meaney MP, John C, Pappan KL, Kinchen JM. Metabolomics-Based Analysis of Banana and Pear Ingestion on Exercise Performance and Recovery. J Proteome Res. 2015 Dec 4;14(12):5367-77. doi: 10.1021/acs.jproteome.5b00909. Epub 2015 Nov 23. PMID 26561314
- [Derived] Nieman DC, Gillitt ND, Chen GY, Zhang Q, Sakaguchi CA, Stephan EH. Carbohydrate intake attenuates post-exercise plasma levels of cytochrome P450-generated oxylipins. PLoS One. 2019 Mar 18;14(3):e0213676. doi: 10.1371/journal.pone.0213676. eCollection 2019. PMID 30883596
- [Derived] Nieman DC, Gillitt ND, Sha W, Esposito D, Ramamoorthy S. Metabolic recovery from heavy exertion following banana compared to sugar beverage or water only ingestion: A randomized, crossover trial. PLoS One. 2018 Mar 22;13(3):e0194843. doi: 10.1371/journal.pone.0194843. eCollection 2018. PMID 29566095